CLINICAL TRIAL: NCT06993298
Title: Development and Effectiveness of the Augmented Reality Physical Ergonomics (ARPE) Training Module for Manual Material Handling Workers: A Quasi-Experimental Study Protocol
Brief Title: ARPE Training for Manual Handling Workers: A Quasi-Experimental Study on Ergonomic Knowledge and Practice
Acronym: ARPE;MMH
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universiti Teknologi Mara (Other)
Responsible Party: Principal Investigator, Fatimah Zahra Binti Norman, Dr, Universiti Teknologi Mara
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: REC/11/2024 [PG/MR/550]
Record Dates: First submitted 2025-05-14; First posted 2025-05-28 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Occupational Diseases; Work Related Upper Limb Disorder
Keywords: Augmented Reality (AR); Ergonomic; Work Related Musculo skeletal Disorder (WMSD)
MeSH Terms: conditions — Occupational Diseases

STUDY DESIGN:
Intervention Model Description: This study uses a quasi-experimental, two-arm, parallel-group design to evaluate the effectiveness of an Augmented Reality Physical Ergonomics (ARPE) training module among manual material handling (MMH) workers. Participants are non-randomly assigned to either the intervention group, which receives ARPE training via the MAKAR XR app, or the control group, which receives conventional ergonomic training based on national DOSH guidelines. The study spans six weeks with assessments at baseline, week 1, and week 6. The primary outcome is ergonomic knowledge, while secondary outcomes include self-prevention and self-evaluation behaviors. Usability of the AR module will also be assessed. This model emphasizes practical workplace relevance and digital health application in occupational training.
Masking Description: This is an open-label study with no masking. Both participants and researchers are aware of group assignments (intervention vs. control). Due to the nature of the intervention-an Augmented Reality training module versus conventional training-it is not feasible to blind participants or outcome assessors.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional Ergonomics Training (Active Comparator): Participants in this arm will undergo conventional ergonomic training based on the Department of Occupational Safety and Health (DOSH) guidelines. The training will be delivered through traditional methods such as lectures, printed materials, and visual presentations. The content includes safe manual handling techniques, identification of work-related musculoskeletal disorder (WMSD) risk factors, and best practices for injury prevention.
  Interventions: Behavioral: Conventional Ergonomics Training
- Augmented Reality Ergonomics Training (Experimental): Participants in this arm will receive an immersive Augmented Reality-based ergonomics training module known as ARPE, delivered through the MAKAR XR mobile application. The training content is aligned with ergonomic guidelines for manual material handling (MMH) tasks and includes 3D interactive simulations, visual demonstrations of proper lifting techniques, and safety practices. The training aims to improve ergonomic knowledge, encourage self-prevention of work-related musculoskeletal disorders (WMSDs), and enhance self-evaluation of posture and manual handling behaviors. The module is self-paced and supported by weekly WhatsApp check-ins throughout the 6-week intervention period.
  Interventions: Device: Augmented Reality Ergonomics Training (ARPE)

INTERVENTIONS:
Device: Augmented Reality Ergonomics Training (ARPE) — Participants in this arm will receive an interactive training module using Augmented Reality (AR) delivered via the MAKAR XR app. The module aims to enhance ergonomic knowledge, self-prevention, and self-evaluation related to work-related musculoskeletal disorders (WMSDs)
  Arms: Augmented Reality Ergonomics Training
Behavioral: Conventional Ergonomics Training — Participants in this arm will receive conventional ergonomic training based on the Department of Occupational Safety and Health (DOSH) guidelines for manual material handling (MMH) workers. The training includes lectures, printed materials, and standard instructional content focused on safe lifting techniques, proper posture, risk factor identification, and strategies to prevent work-related musculoskeletal disorders (WMSDs). This training is delivered in a one-time session with follow-up reminders, simulating current standard practices in workplace safety education.
  Arms: Conventional Ergonomics Training

SUMMARY:
The goal of this study is to evaluate whether an Augmented Reality-based ergonomic training module (ARPE) can improve ergonomic knowledge, self-prevention, and self-evaluation practices among adult manual material handling (MMH) workers in warehouses. The main questions it aims to answer are:

Does the ARPE training module improve workers' ergonomic knowledge?

Does it enhance their ability to prevent and assess risks of work-related musculoskeletal disorders (WMSDs)?

Researchers will compare an intervention group using the ARPE module with a control group receiving traditional training based on national ergonomic guidelines to see if the AR module leads to better outcomes.

Participants will:

Attend a briefing and use the ARPE training via the MAKAR XR app

Complete self-assessment questionnaires at baseline, week 1, and week 6

Receive reminders and follow-ups through WhatsApp

DETAILED DESCRIPTION:
This study is a quasi-experimental trial designed to develop and evaluate the effectiveness of the Augmented Reality Physical Ergonomics (ARPE) training module among manual material handling (MMH) workers in Malaysia. MMH workers face a high risk of developing work-related musculoskeletal disorders (WMSDs) due to frequent lifting, carrying, and handling of heavy objects. Traditional ergonomic training methods-such as lectures and printed materials-have been found to be less engaging and may not lead to effective behavior change.

The ARPE module uses Augmented Reality (AR) technology through the MAKAR XR mobile app to provide immersive and interactive ergonomic training. The goal is to enhance the understanding of proper manual handling techniques, promote self-assessment, and encourage preventive behaviors in real work settings.

Two groups will be included in the study:

Intervention group: receives ARPE training using the MAKAR XR app

Control group: receives conventional ergonomic training based on national DOSH (Department of Occupational Safety and Health) guidelines

The study includes three phases:

Introduction phase: Participants are briefed on their training, and baseline data is collected on ergonomic knowledge and practices.

Intervention phase: Participants interact with their respective training (ARPE or conventional), with engagement monitored and supported via WhatsApp.

Post-intervention phase (6 weeks later): Participants complete follow-up questionnaires to assess retention of ergonomic knowledge and application of safe practices.

The main outcomes are improvement in ergonomic knowledge (primary), and changes in self-prevention and self-evaluation behaviors (secondary). Usability of the ARPE module will also be assessed using a validated mobile health app questionnaire (M-MAUQ).

This study aims to demonstrate that AR-based training can be a more effective and engaging alternative to traditional methods, potentially reducing the risk of WMSDs and improving workplace safety.

ELIGIBILITY:
Inclusion Criteria:

Malaysian citizen

Age 18 years and above

Currently employed as a manual material handling (MMH) worker in a warehouse

Regularly performs MMH tasks (e.g., lifting, lowering, pushing, pulling, carrying, holding, or restraining objects weighing 14 kg or more)

Works a minimum of 8 hours per day in a role involving MMH

Owns a mobile phone capable of downloading and running the MAKAR XR app

Exclusion Criteria:

Pregnant

Currently an intern or temporary worker

Has undergone ergonomic training within the past six months

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 78 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Improvement in Ergonomic Knowledge | Baseline (T0) - Prior to training Week 1 Post-Training (T1) Week 6 Follow-Up (T6)
  Description:
  Participants' ergonomic knowledge will be assessed using the Ergonomic Knowledge Domain Questionnaire, a validated 8-item multiple-choice instrument measuring understanding of ergonomic principles, awareness of risk factors for work-related musculoskeletal disorders (WMSDs), and correct manual handling practices.
  Scale Title: Ergonomic Knowledge Domain Questionnaire
  Score Range: 0 to 8
  Scoring: 1 point per correct answer
  Interpretation:
  0-3 = Low knowledge
  4-5 = Moderate knowledge
  6-8 = High knowledge
  Outcome Direction: Higher scores reflect improved ergonomic knowledge and better learning outcomes following the ARPE training module.
  The effectiveness of the intervention will be determined by comparing the scores across three time points between the intervention and control groups.

SECONDARY OUTCOMES:
Improvement in Self-Prevention Practices Toward Ergonomic Risks | Baseline (T0) - Prior to training Week 1 Post-Training (T1) Week 6 Follow-Up (T6)
  This outcome will be measured using the Self-Prevention Domain Questionnaire, a validated 6-item self-assessment instrument using a 7-point Likert scale to evaluate participants' self-reported preventive behaviors and attitudes toward managing ergonomic risks at the workplace.
  Scale Title: Self-Prevention Domain Questionnaire
  Score Range: 6 to 42
  Scoring: Each item is rated from 1 (Strongly Disagree) to 7 (Strongly Agree)
  Interpretation:
  6-21 = Poor self-prevention
  22-31 = Moderate self-prevention
  32-42 = Good self-prevention
  Outcome Direction: Higher scores indicate greater awareness and better self-preventive ergonomic practices.
  Scores will be compared between the intervention and control groups at three assessment points to determine changes in prevention practices after training.

OTHER OUTCOMES:
Improvement in Self-Evaluation of Ergonomic Practices | Baseline (T0) - Prior to training Week 1 Post-Training (T1) Week 6 Follow-Up (T6)
  This outcome will be measured using the Self-Evaluation Domain Questionnaire, a validated 5-item instrument using a 7-point Likert scale to assess how frequently participants apply ergonomic principles in their daily work practices and reflect on their own ergonomic behavior following the training.
  Scale Title: Self-Evaluation Domain Questionnaire
  Score Range: 5 to 35
  Scoring: Each item is rated from 1 (Never) to 7 (Always)
  Interpretation:
  5-17 = Low ergonomic self-practice
  18-26 = Moderate ergonomic self-practice
  27-35 = High ergonomic self-practice
  Outcome Direction: Higher scores indicate more frequent application and internalization of ergonomic practices, reflecting the participant's behavioral response to the training.
  Scores will be compared between the intervention and control groups at three time points to assess sustained behavioral changes.

REFERENCES:
- [Derived] Norman FZ, Yasin SM, Mohamad M, Azzani M. Augmented Reality Physical Ergonomics (ARPE) Training for Manual Material Handling Workers: A Protocol for a Quasi-experimental Study. Cureus. 2025 Sep 14;17(9):e92302. doi: 10.7759/cureus.92302. eCollection 2025 Sep. PMID 41111705